CLINICAL TRIAL: NCT01903694
Title: Randomized Trial Sorafenib-Pravastatin Versus Sorafenib Alone for the Palliative Treatment of Child-Pugh A Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JOUVE PHRC K 2009
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Child-Pugh A Hepatocellular Carcinoma
MeSH Terms: interventions — Sorafenib; Pravastatin

ARMS (2):
- sorafenib (Active Comparator): 800 mg of sorafenib twice daily orally.
  Interventions: Drug: Sorafenib
- sorafenib-pravastatin (Experimental): 800 mg of sorafenib twice daily oral doses associated with 40 mg of pravastatin in a taken per os. Pravastatin will be taken during dinner.
  Interventions: Drug: Sorafenib + Pravastatin

INTERVENTIONS:
Drug: Sorafenib + Pravastatin
  Other Names: 800 mg of sorafenib twice daily oral doses associated with; 40 mg of pravastatin in a taken per os. Pravastatin will be taken during dinner.
  Arms: sorafenib-pravastatin
Drug: Sorafenib
  Other Names: 800 mg of sorafenib twice daily orally.
  Arms: sorafenib

SUMMARY:
Principal objective: to evaluate the effect of the combination pravastatin - sorafenib versus sorafenib alone on overall survival in patients with hepatocellular carcinoma developing on Child-Pugh A cirrhosis who are unsuitable for curative treatment.

Secondary objectives: evaluate the effect of this treatment on progression-free survival, the time to progression, the time to treatment failure and quality of life (QLQ-C30 et FACT HEP)

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma diagnosed by:
* either a histological examination
* or if histological evidence cannot be obtained (ascites, coagulation disorders) the diagnosis can be made in cases of cirrhosis according to EASL/AASLD 2005 criteria, by revealing a hepatic focal lesion of more than 10 mm
* on two dynamic imaging techniques (helical CT-scan, MRI, contrast-enhanced ultrasound) for tumours measuring less than 2 cm. The lesion must be characterised by hyperdensity during the arterial phase and wash-out during the delayed portal phase Patients who are not suitable for treatment with a curative intent (transplantation, resection, percutaneous destruction) or by chemo-embolisation or with progressive hepatocellular carcinoma after the failure of specific treatment Prognostic CLIP score 0 to 4 Child-Pugh Class A Transaminases ≤ 5 N and Creatininemia ≤ 1.5 N WHO: 0, 1 or 2 Age more than 18 years Foreseeable survival > 12 weeks Possibility of regular follow-up Written informed consent

Exclusion Criteria:

* Extra-hepatic disease that could be life-threatening in the short or medium term Another progressive cancer with the exception of in situ cervical cancer, a superficial bladder tumour and treated basocellular carcinoma.

Any other cancer treated with a curative intent in the previous 3 years can be included in the study Heart failure (≥New York Heart Association class 2), uncontrolled AHT or arrhythmia, myocardial infarction in the previous 6 months Digestive haemorrhage in the previous month Patients who are receiving or have already received treatment with statins or sorafenib Pregnancy and breast-feeding. Women of child-bearing age must use an effective method of contraception throughout the trial and for 3 months after the end of the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
determination of the tumor according to the evaluation criteria of Response Evaluation Criteria in Solid Tumors | To be done within the month preceding baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France

REFERENCES:
- [Result] Jouve JL, Lecomte T, Bouche O, Barbier E, Khemissa Akouz F, Riachi G, Nguyen Khac E, Ollivier-Hourmand I, Debette-Gratien M, Faroux R, Villing AL, Vergniol J, Ramee JF, Bronowicki JP, Seitz JF, Legoux JL, Denis J, Manfredi S, Phelip JM; PRODIGE-11 investigators/collaborators. Pravastatin combination with sorafenib does not improve survival in advanced hepatocellular carcinoma. J Hepatol. 2019 Sep;71(3):516-522. doi: 10.1016/j.jhep.2019.04.021. Epub 2019 May 22. PMID 31125576